CLINICAL TRIAL: NCT03768765
Title: Duration of Medication Therapy and Outcomes After Holmium Laser Prostate Surgery for Patients With Benign Prostatic Hyperplasia (BPH)
Status: Terminated | Type: Observational
Why Stopped: Slow recruitment of patients who have been on medication for under a year for benign prostatic hyperplasia
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Don Neff, MD, FACS, Associate Professor, University of Kansas Medical Center
Other Study IDs: 143049
Record Dates: First submitted 2018-12-03; First posted 2018-12-07 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Long Term Medication Usage: Patients who have been on medication for over a year for benign prostatic hyperplasia (BPH)
  Interventions: Procedure: Holmium Laser Prostate Surgery
- Short Term Medication Usage: Patients who have been on medication for under a year for benign prostatic hyperplasia (BPH)
  Interventions: Procedure: Holmium Laser Prostate Surgery

INTERVENTIONS:
Procedure: Holmium Laser Prostate Surgery — Patients will undergo standard of care holmium laser prostate surgery

SUMMARY:
To determine if the prior prolonged use of medication, as a treatment for benign prostatic hyperplasia, reduces the efficacy of Holmium laser enucleation of the prostate (HoLEP) for patients with benign prostatic hyperplasia (BPH).

DETAILED DESCRIPTION:
Experience from clinic has suggested that men who receive medication for long periods of time, defined as over a year for study purposes, have a poorer response to surgical treatment for benign prostatic hyperplasia (BPH). It has previously been demonstrated that medication use does not alter the perioperative outcomes after HoLEP; however, to our knowledge, no study to date has investigated holmium laser prostate surgery outcomes associated with the duration of pre-operative medication therapy.

Some of the more common medications for BPH are alpha-1 blockers and 5-alpha-reductase inhibitors. A five-year study of patients showed that treatment failure, defined as need for surgery or conversion to other medication, was observed in 18.8% of patients who were prescribed tamsulosin, an alpha-1 blocker, for BPH. The study further suggested that treatment with this class of medication may not be appropriate long-term for those patients with a large prostate volume and/or a large post-void residual volume. Similar results have been demonstrated with 5-alpha-reductase inhibitors, with more than 30% of men not responding to its therapeutic effects.

The progression of BPH symptoms is complex and the result of multiple pathways such as androgen receptor signaling, proinflammatory cytokines, and growth factor signals, all of which can be affected by medication. 5-alpha-reductase inhibitors work by limiting the conversion of testosterone to dihydrotestosterone. An overabundance of dihydrotestosterone can affect the regulation of cell cycle, cell growth, and differentiation in the prostate, leading to BPH. Alpha-1 blockers work by mediating prostate smooth-muscle relaxation though it is unclear if this specific action is the reason for the relief of BPH symptoms. Considering the aforementioned pathways, the goal of this clinical trial is to investigate if a prolonged period of medication is associated with the effectiveness of holmium laser surgery. By grouping patients based on medication treatment time, the goal is to determine if their responses are different and clinically significant, in order to better inform standard of care practices for those with BPH.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 18 years of age or older
2. Patients must present to clinic with a diagnosis of benign prostatic hyperplasia with lower urinary tract symptoms
3. Patients must be scheduled to undergo a holmium laser prostate surgery (enucleation or ablation)

Exclusion Criteria:

1. Patients who are under 18 years of age are not eligible.
2. Patients who have a diagnosis of bladder cancer are not eligible.
3. Patient who have a diagnosis of prostate cancer are not eligible.
4. Patients with an elevated prostate-specific antigen (PSA) suggesting prostate cancer are not eligible unless patient has prior negative prostate biopsy.
5. Patients who have acute prostatitis, a prostate abscess, or neurogenic bladder are not eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will present to clinic for treatment of BPH
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2024-08-27 (Actual)

PRIMARY OUTCOMES:
Bladder Function | Six Months
  The primary objective is to determine if patients who undergo holmium laser surgery prior to being placed on long term medication for benign prostatic hyperplasia (BPH) have a greater improvement in their bladder function, as measured by urodynamics, when compared to patients who undergo holmium laser surgery after being placed on long term medication for BPH.

SECONDARY OUTCOMES:
Improvement in Quality of Life | Six Months
  The secondary objectives are to determine if patients who undergo holmium laser surgery prior to long term medication for benign prostatic hyperplasia (BPH) have a greater improvement in their quality of life, as measured by questionnaires, when compared to patients who under holmium laser surgery after having received long term medication.
Complete Emptying | Six Months
  The secondary objectives are to determine if patients who undergo holmium laser surgery prior to long term medication for benign prostatic hyperplasia have great improvement in complete emptying of their bladder, as measured by post void residual volume (PVR), when compared to patients who under holmium laser surgery after having received long term medication.
Lower Urinary Tract Symptoms | Six Months
  The secondary objectives are to determine if patients who undergo holmium laser surgery prior to long term medication for benign prostatic hyperplasia have great improvement in regards to their lower urinary tract symptoms, as measured by the American Urology Association (AUA) symptom score, when compared to patients who under holmium laser surgery after having received long term medication. The AUA symptom score is a measure of lower urinary tract symptoms and is scored on a scale of 0-25, with a score in the range of 0-8 indicating mild symptoms, 9-19 indicating moderate symptoms, and a score in 20-35 range indicating severe symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Health System, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No